CLINICAL TRIAL: NCT04014868
Title: During-exercise Physiological Effects of Nasal High-flow in Patients With Chronic Obstructive Pulmonary Disease
Acronym: AIRVO-PHYSIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ADIR Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AIRVO-PHYSIO
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; Exercise; Nasal high flow; Muscle
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Intervention Model Description: Single-blind randomized cross-over study.
Who Masked: Participant
Masking Description: The nasal high-flow device will be out of sight of the patients and will not be switched ON. The oxygen connection at the exit of the device will be obstructed. If the patient needs supplementary oxygen during-exercise, it will be provided through the fitting located just before the nasal canula (see Arms, Experimental: Nasal high-flow).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasal high-flow (Experimental): Patients will perform a constant workload exercise testing (75% of the maximal workload achieved during a previously performed incremental cardiopulmonary exercise testing) with active nasal high-flow :
  Flow : 30 L/min; Temperature : 34°C;
  The device will be out of sight of the patient. The device allow for oxygen supplementation (fitting on the back of the device). Usual oxygen prescription (if any) will be adjusted to reach a transcutaneous oxygen saturation superior to 90%. A second fitting will be placed just before the nasal canula to allow for oxygen supplementation during the sham nasal high-flow (device turned OFF) test.
  Due to the cross-over design of the study, all patients will perform both interventions.
  Interventions: Device: Nasal high-flow
- Sham nasal high-flow (Sham Comparator): Patients will perform a constant workload exercise testing (75% of the maximal workload achieved during a previously performed incremental cardiopulmonary exercise testing) with a sham nasal high-flow :
  The procedure will be exactly the same but the device (out of sight of the patient) will be turned OFF. Oxygen supplementation will be possible through the fitting placed just before the nasal canula.
  Due to the cross-over design of the study, all patients will perform both interventions.
  Interventions: Other: Sham nasal high-flow

INTERVENTIONS:
Device: Nasal high-flow — See arm description.
  Arms: Nasal high-flow
Other: Sham nasal high-flow — See arm description.
  Arms: Sham nasal high-flow

SUMMARY:
Chronic obstructive pulmonary disease is a major cause of disability and mortality worldwide. This disease progressively leads to dyspnea and exercise capacity impairment. Pulmonary rehabilitation teaches chronic obstructive pulmonary disease patients to cope effectively with the systemic effects of the disease and improves exercise capacity, dyspnea and quality of life in patients with chronic obstructive pulmonary disease. However, the best training modality remains unknown. Physiological studies highlight the benefit of high intensity endurance training. However, many patients do not tolerate such a training due to ventilatory limitation and dyspnea. Therefore, a strategy to reduce dyspnea would allow a greater physiological muscle solicitation and improvement. Thus, many studies focus on means to increase exercise tolerance in patients with chronic obstructive pulmonary disease.

Nasal high flow delivers heated and humidified high flow air (up to 60 L/min) through nasal cannula providing physiological benefits such as positive airway pressure and carbon dioxide washout. It can be used in association with oxygen and offers the advantage to overtake the patient's inspiratory flow, providing a stable inspired fraction of oxygen. Nasal high flow has widely been studied in pediatric and adult intensive care units and seems better than conventional oxygen therapy and as effective as noninvasive ventilation with regards to mortality to treat hypoxemic acute respiratory failure.

More recently, nasal-high flow has been shown to improve endurance exercise capacity in patients with chronic obstructive pulmonary disease. However, the underlying physiological mechanisms have not been yet elucidated but may help to optimise the utilization of the device.

Therefore, the primary objective of this study is to assess the respiratory physiological effects nasal high-flow during-exercise in stable patients with chronic obstructive pulmonary disease.

Secondary objectives are to assess the effects nasal high-flow during-exercise on endurance capacity, respiratory drive, dynamic hyperinflation, cardiorespiratory pattern and muscular metabolism.

DETAILED DESCRIPTION:
Experimental design:

Patients referred for pulmonary rehabilitation will be approached to participate in this study. Eligible patients who agree to participate in the study and sign informed consent will perform two constant workload exercise testing the same day with either nasal high-flow or sham nasal high-flow (separated by a 1 hour rest-period) in a randomized order.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18years and < 80years;
* Chronic obstructive pulmonary disease Gold III-IV;
* Stable (no exacerbation) in the past 4 weeks;
* Referred for pulmonary rehabilitation (no cardiac, neurological, orthopedic, neuromuscular, psychological or psychiatric contra indication).

Non-inclusion Criteria:

* Acute exacerbation of chronic obstructive pulmonary disease between the incremental cardiopulmonary exercise testing and inclusion;
* Tracheostomy;
* Nasal high flow intolerance;
* Pregnancy or likely to be;
* Unable to consent;
* Patients under guardianship.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-10 (Actual)

PRIMARY OUTCOMES:
Transdiaphragmatic pressure-time product using a single-use catheter with two balloons to measure gastric and esophageal pressures. | The outcome will be continuously recorded during the two constant workload exercise testing. The 2 tests will be performed the same day for a total time frame of 3hours.
  Transdiaphragmatic pressure is calculated as gastric pressure minus oesophageal pressure. The outcome will be continuously recorded during the two constant workload exercise testing. Results will be shown at time limit and iso time (defined as time limit of the shortest test).

SECONDARY OUTCOMES:
Ventilatory drive using diaphragmatic electromyogram through the same single-use catheter used for transdiaphragmatic pressure (which is provided with 6 pairs of electrodes). | The outcome will be continuously recorded during the two constant workload exercise testing. The 2 tests will be performed the same day for a total time frame of 3hours.
  Diaphragmatic electromyography will be recorded with 6 pairs of electrodes and will be used as a surrogate for ventilatory drive. Results will be shown at time limit and iso time (defined as time limit of the shortest test).
Ventilatory efficiency using indirect calorimetry | The outcome will be continuously recorded during the two constant workload exercise testing. The 2 tests will be performed the same day for a total time frame of 3hours.
  Ventilatory efficiency will be assessed as the ratio between exercise ventilation to carbon dioxide production. Results will be shown at time limit and iso time (defined as time limit of the shortest test).
Dynamic hyperinflation using the fall in during-exercise inspiratory capacity | The outcome will be recorded during the two tests. The 2 tests will be performed the same day for a total time frame of 3hours.
  Maximal inspiratory maneuver will be performed every minute during the two constant workload exercise testing. Results will be shown at time limit and iso time (defined as time limit of the shortest test).
Transcutaneous arterial carbon dioxide partial pressure using capnography. | The outcome will be continuously recorded during the two constant workload exercise testing. The 2 tests will be performed the same day for a total time frame of 3hours.
  The outcome will be measured at the earlobe. Results will be shown at time limit and iso time (defined as time limit of the shortest test).
Dyspnea during the constant workload exercise testing using modified Borg scale (0-10). | The outcome will be recorded during the two tests. The 2 tests will be performed the same day for a total time frame of 3hours.
  Borg scale range from 0 (no breathlessness) to 10 (maximal breathlessness). The dyspnea will be assessed every 30sec during the constant workload exercise testing. Results will be shown at time limit and iso time (defined as time limit of the shortest test).
Vastus lateralis muscle peripheral perfusion during exercise using near infrared spectroscopy. | The outcome will be recorded during the two tests. The 2 tests will be performed the same day for a total time frame of 3hours.
  The outcome will be assessed every minute. Peripheral muscle perfusion will be assessed using the linear increase in total haemoglobin and myoglobin during a venous occlusion (20 seconds) and used as a surrogate for local blood perfusion. Results will be shown at time limit and iso time (defined as time limit of the shortest test).
Vastus lateralis muscular peripheral oxygen extraction during exercise using near infrared spectroscopy. | The outcome will be recorded during the two tests. The 2 tests will be performed the same day for a total time frame of 3hours.
  The outcome will be assessed continuously. Vastus lateralis muscle oxygen extraction will be assessed using deoxyhaemoglobin and deoxymyoglobin as a surrogate for peripheral oxygen extraction. Results will be shown at time limit and iso time (defined as time limit of the shortest test).
Endurance exercise capacity in seconds. | The outcome will be measured after every test. Data will be continuously collected during the tests. The 2 tests will be performed the same day for a total time frame of 3hours.
  Patients will perform a constant workload exercise testing at 75% of the maximal workload achieved during the incremental cardiopulmonary exercise testing.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Cuvelier, MD, PhD, Prof, Principal Investigator — Normandie University, UNIROUEN, UPRES EA 3830, Haute Normandie Research and Biomedical Innovation, Rouen, France ; Pulmonary, Thoracic Oncology and Respiratory Intensive Care Department, Rouen University Hospital, Rouen, France; Jean-François Muir, MD, Prof, Study Chair — ADIR Association, Rouen University Hospital, Rouen, France ; Normandie University, UNIROUEN, UPRES EA 3830, Haute Normandie Research and Biomedical Innovation, Rouen, France; Maxime Patout, MD, Msc, Study Chair — Normandie University, UNIROUEN, UPRES EA 3830, Haute Normandie Research and Biomedical Innovation, Rouen, France ; Pulmonary, Thoracic Oncology and Respiratory Intensive Care Department, Rouen University Hospital, Rouen, France; Tristan Bonnevie, Msc, Study Chair — UADIR Association, Rouen University Hospital, Rouen, France ; niversity, UNIROUEN, UPRES EA 3830, Haute Normandie Research and Biomedical Innovation, Rouen, France; Francis-Edouard Gravier, Msc, Study Chair — ADIR Association, Rouen University Hospital, Rouen, France ; Normandie University, UNIROUEN, UPRES EA 3830, Haute Normandie Research and Biomedical Innovation, Rouen, France
Locations (1):
- ADIR Association, Bois-Guillaume, France